CLINICAL TRIAL: NCT06087926
Title: Investigation of Non-invasive Brain Stimulation for the Treatment of Apathy
Brief Title: Apathy in Parkinson Disease TMS Study
Acronym: PDTMSAPATHY
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 23-1829; K23MH132884 (NIH)
Record Dates: First submitted 2023-10-11; First posted 2023-10-18 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-05

CONDITIONS: Parkinson Disease
Keywords: Apathy; Motivation
MeSH Terms: conditions — Parkinson Disease; Lethargy | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participant will be blinded as to which site is being stimulated, experimental site or control site.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Medial Prefrontal Cortex - Control Site (Experimental): Participants first undergo transcranial magnetic stimulation to the medial prefrontal cortex. After a 3-week washout period, participants then undergo transcranial magnetic stimulation to the control site.
  Interventions: Device: Transcranial Magnetic Stimulation (TMS)
- Control Site - Medial Prefrontal Cortex (Experimental): Participants first undergo transcranial magnetic stimulation to the control site. After a 3-week washout period, participants then undergo transcranial magnetic stimulation to the medial prefrontal cortex.
  Interventions: Device: Transcranial Magnetic Stimulation (TMS)

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation (TMS) — Transcranial magnetic stimulation (or TMS) is a non-invasive form of brain stimulation in which a magnetic pulse is applied directly to the scalp. TMS is FDA approved for the treatment of depression and other neuropsychiatric disorders and is regularly used in neurologic and psychiatric research.
  ITBS is a particular TMS protocol which delivers the magnetic field in triplet bursts (three stimulations very close together at a frequency of 50 Hz). The triplet bursts are repeated at a rate of 5 Hz for 2 seconds (30 pulses), followed by 8 seconds rest, repeated 20 times for a total of 600 pulses. Each treatment lasts approximately 3 minutes.
  Other Names: Intermittent Theta-Burst Stimulation (iTBS)

SUMMARY:
The goal of this clinical trial is to develop non-invasive brain stimulation targets for the treatment of apathy, or motivation problems, in Parkinson Disease.

The main questions the study aims to answer are:

1. Does transcranial magnetic stimulation change effort task performance in Parkinson's Disease patients?
2. Is there a link between brain signals and apathy?

Participants will

* complete questionnaires and assessments
* perform an effort task
* have their brain activity recorded (EEG)
* receive non-invasive brain stimulation (TMS)

Researchers will compare two stimulation locations (experimental site and control site) to see if TMS of the experimental site has an effect on apathy. Participants will receive stimulation of both sites (during separate visits).

DETAILED DESCRIPTION:
Participants will be asked to come for 3 study visits.

During visit 1, after being informed about the study and potential risks, all patients giving written informed consent will undergo a brief cognitive assessment, a movement examination, and answer questionnaires. Additionally, the individual motor threshold will be determined for each participant. Visit 1 will take 2-3 hours.

Visits 2 and 3 will involve:

* completing questionnaires,
* performing a task where fictitious rewards can be earned by squeezing a dynamometer,
* recording brain activity with an electroencephalogram (EEG), and
* receiving transcranial magnetic stimulation (TMS). Visits 2 and 3 will take approximately 3 hours each and will be separated from each other by at least 3 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of idiopathic Parkinson Disease.
* At least 5 years of symptoms.
* On dopaminergic medication for Parkinson Disease.
* Stable on dopaminergic medication and other medications which may influence apathy (such as selective serotonin re-uptake inhibitors, stimulant medications) for at least 4 weeks prior to first study visit and remain stable throughout the study period.
* Hospital's study-specific informed consent must be obtained.
* Must have capacity to provide informed consent in English.
* For female participants, confirmation that they have not had a menstrual period in over 12 months, or that they will use an effective form of contraception during the study.

Exclusion Criteria:

* Inability to provide informed consent.
* Inability to perform effort task (determined during the titration session).
* Presence of dementia (Montreal Cognitive Assessment (MoCA) score < 21).
* History of epilepsy or brain surgery.
* Severe tremor or dyskinesia that would interfere with EEG (determined by the PI).
* Patients with clinically significant medical or neurological conditions which may be an alternative cause of parkinsonism such as repeated brain injury, anti-dopaminergic medications, anoxic brain injury, or significant basal ganglia strokes.
* Presence of other known central nervous system disease that may interfere with performance or interpretation of EEG or TMS.
* Presence of any implanted metal devices including, but not limited to, pacemakers, deep brain stimulators, vagal nerve stimulators, bladder stimulators, or cochlear implants.
* Presence of medical contraindications to TMS such as implanted stimulators, history of mania or bipolar disorder, history of epilepsy.

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in goal-directed behavior after transcranial magnetic stimulation (TMS) | Immediately before stimulation and 15 minutes after stimulation.
  Differences in the degree of change in goal-directed behavior after brain stimulation at each site (medial prefrontal cortex or control site).
  Goal-directed behavior will be determined using the streamlined version of the Expenditure of Effort for Reward Task (S-EEfRT). In the S-EEfRT, participants choose to complete either a "Hard" task or an "Easy" task for variable monetary incentives.
Change in reward evaluation after transcranial magnetic stimulation (TMS) | Immediately before stimulation and 15 minutes after stimulation.
  Differences in the degree of change in reward evaluation after brain stimulation at each site (medial prefrontal cortex or control site).
  Reward evaluation will be determined using the streamlined version of the Expenditure of Effort for Reward Task (S-EEfRT). In the S-EEfRT, participants choose to complete either a "Hard" task or an "Easy" task for variable monetary incentives.

SECONDARY OUTCOMES:
Association between frontal midline theta EEG power and goal-oriented behavior | Approximately 45 minutes before and 45 minutes after stimulation.
  Degree of association between frontal midline theta EEG power and goal-oriented behavior.
  Goal-directed behavior will be determined using the streamlined version of the Expenditure of Effort for Reward Task (S-EEfRT). In the S-EEfRT, participants choose to complete either a "Hard" task or an "Easy" task for variable monetary incentives.
Association between frontal midline theta EEG power and reward evaluation | Approximately 45 minutes before and 45 minutes after stimulation.
  Degree of association between frontal midline theta EEG power and reward evaluation.
  Reward evaluation will be determined using the streamlined version of the Expenditure of Effort for Reward Task (S-EEfRT). In the S-EEfRT, participants choose to complete either a "Hard" task or an "Easy" task for variable monetary incentives.

OTHER OUTCOMES:
Association between frontal midline theta EEG power and subjective apathy | Approximately 45 minutes before and 45 minutes after stimulation.
  Degree of association between frontal midline theta EEG power and subjective apathy as measured with the Lille Apathy Rating Scale (LARS).
  The LARS has been validated in Parkinson Disease. It consists of a structured interview that includes 33 items. Responses are scored on a dichotomous scale. The LARS score will be investigated as an effect measure modifier in the association between performance on the S-EEfRT and frontal midline theta power.

CONTACTS AND LOCATIONS:
Overall Officials: Miriam Sklerov, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- UNC-Chapel Hill, Cassidy Lab, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Supporting Information: Study Protocol
Time Frame: Beginning 9 and continuing for 36 months after publication.
Access Criteria: Data will be made available to investigators who have approval from an IRB, IEC, or REB and an executed data use/sharing agreement with UNC.